CLINICAL TRIAL: NCT04045964
Title: Nicotine Patch as an Adjunctive Intervention to Reduce Secondhand Smoke Among NICU Families
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Angela L Stotts, Professor and Vice Chair for Research (Department of Family & Community Medicine), The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-11-0641(Substudy)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Results first posted 2019-09-17 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2019-10

CONDITIONS: Environmental Tobacco Smoke; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational advice and free NRT (Experimental)
  Interventions: Drug: nicotine replacement therapy (NRT); Behavioral: motivational advice
- Quitline referral (Active Comparator)
  Interventions: Behavioral: Quitline referral

INTERVENTIONS:
Drug: nicotine replacement therapy (NRT) — Participants were provided with either 2 weeks of 14-mg or 21-mg transdermal nicotine patches for every smoker in the home
  Other Names: nicotine patch
  Arms: Motivational advice and free NRT
Behavioral: motivational advice — Received two in-hospital motivational advice sessions by a research associate (RA). The RA adapted session content from a previous tobacco-smoke exposure protocol
  Arms: Motivational advice and free NRT
Behavioral: Quitline referral — Quitline participants received information about tobacco-smoke exposure reduction and a referral to a tobacco Quitline.
  Arms: Quitline referral

SUMMARY:
The purpose of this study was to explore the potential for directly targeting smoking cessation, regardless of motivation level, in a subsample of neonatal intensive care unit (NICU) parents with the ultimate goal of reducing secondhand smoke (SHS) in their homes.

ELIGIBILITY:
Inclusion Criteria:

* Eligible mothers of any age or ethnic background must have an infant that is at least 1 week prior to the estimated date of hospital discharge in the NICU (ensuring time for the intervention)
* report that a household resident smokes at least 5 cigarettes per day, on average, within the 2 months preceding the screening visit
* agree to attend intervention sessions
* live within 50 miles of our center
* and have access to a telephone

Exclusion Criteria:

* Mothers were ineligible if they met criteria for severe cognitive, and/or psychiatric impairment, per judgment of NICU and research staff, that precludes cooperation with study protocol
* were unable to read, write, and speak English
* were unable or unwilling to provide signed consent for participation
* and were unable or unwilling to meet study requirements for data collection and intervention purposes.
* Within the month immediately preceding the screening visit, use of any form of tobacco or nicotine products other than cigarettes (e.g., e-cigarettes, chewing tobacco, etc.) on 3 or more days within a week if the individual refuses to refrain from such tobacco use during the course of the study
* Current use of NRT or enrollment (or plans to enroll) in another smoking cessation program in the next 3 months
* Uncontrolled hypertension (systolic blood pressure [SBP] greater than 180 or diastolic blood pressure [DBP] greater than 110)
* History of severe cardiovascular (stroke, heart attack), kidney (e.g. chronic or acute kidney failure) or liver disease, or other unstable disease in the last 3 months
* History of hypersensitivity or allergic reaction to NRT or similar chemical classes or any component of these formulations (including allergy to latex)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-29 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela L Stotts, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Advice and Free NRT: nicotine replacement therapy (NRT): Participants were provided with 2 weeks of either 14-mg or 21-mg transdermal nicotine patches for every smoker in the home
  motivational advice: Received two in-hospital motivational advice sessions by a research associate (RA).
Period: Overall Study
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Started | 16 | 16
Intervention Visit(s) | 15 | 16
Follow up Visit 1 | 15 | 15
Follow up Visit 2 | 15 | 15
Completed | 15 | 15
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Advice and Free NRT | Quitline Referral | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (9.7) | 29.9 (4.3) | 30.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African-America | 9 | 9 | 18
  White, non-Hispanic | 3 | 4 | 7
  Hispanic | 3 | 2 | 5
  Asian | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Number of Participants Who Accepted NRT Patches From Research Staff.
Time Frame: From time of randomization to intervention session number 2 (generally completed within 2-3 weeks of randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT
Number analyzed (Participants) | 16
Participants | 13

2. Primary Outcome: Efficacy as Assessed by the Number of Participants Who Reported That Anyone in Their Household Used NRT.
Time Frame: From time of randomization to follow-up visit #2 (generally completed within 2-3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 16 | 16
Participants | 6 | 2

3. Secondary Outcome: Cigarette Use (Point Prevalence), as Measured by Number of Cigarettes Smoked Per Day by the Participant
Time Frame: Baseline
Population: Only current smokers (at Baseline) were assessed on this measure; 2 reported current smoking (Motivational Advice and Free NRT arm); 3 reported current smoking (Quitline Referral arm). A 4th Quitline participant began smoking after data were collected; therefore, number of cigarettes/day at baseline was not collected for this 4th participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 2 | 3
Participants
  <10 cigarettes per day | 2 | 2
  >=10 cigarettes per day | 0 | 1

4. Secondary Outcome: Cigarette Use (Point Prevalence), as Measured by Number of Cigarettes Smoked Per Day by the Participant's Partner
Time Frame: baseline
Population: Only current smokers were assessed for this measure. 12 partners of participants in the Motivational Advice and Free NRT arm reported current smoking, and 12 partners of participants in the Quitline Referral arm reported current smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 12 | 12
Participants
  <10 cigarettes per day | 6 | 7
  >=10 cigarettes per day | 6 | 5

5. Secondary Outcome: Cigarette Use (Point Prevalence), as Measured by Number of Cigarettes Smoked Per Day by Other Household Members (Other Than the Participant or Participant's Partner)
Time Frame: baseline
Population: Only current smokers were assessed for this measure. 7 household members (other than participant or partner) living with participant in the Motivational Advice and Free NRT arm reported current smoking, and 6 household members (other than participant or partner) living with participant in the Quitline Referral arm reported current smoking.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 7 | 6
Participants
  <10 cigarettes per day | 5 | 3
  >=10 cigarettes per day | 2 | 3

6. Secondary Outcome: Smoking Quit Attempts, as Measured by Number of Participants Who Reported One or Greater Quit Attempts
Time Frame: at the time of follow-up visit #1 (about 2 weeks post-intervention)
Population: Only participants who reported current smoking were assessed for this measure. 2 participants in the Motivational Advice and Free NRT arm reported current smoking, and 4 participants in the Quitline Referral arm reported current smoking (between baseline and the follow-up visit #1; i.e., 1 Quitline participant began smoking after baseline).
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 2 | 4
Participants | 2 | 1

7. Secondary Outcome: Smoking Quit Attempts, as Measured by Number of Participants Who Reported One or Greater Quit Attempts
Time Frame: at the time of follow-up visit #2 (about 1 month post-intervention)
Population: Only participants who reported current smoking were assessed for this measure. 2 participants in the Motivational Advice and Free NRT arm reported current smoking, and 4 participants in the Quitline Referral arm reported current smoking (between baseline and the follow-up visit #2; i.e., 1 Quitline participant began smoking after baseline).
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 2 | 4
Participants | 1 | 4

8. Secondary Outcome: Smoking Quit Attempts, as Measured by Number of Participant's Partners Who Reported One or Greater Quit Attempts
Time Frame: at the time of follow-up visit #1 (about 2 weeks post-intervention)
Population: For each arm, 12 partners reported current smoking at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 12 | 12
Participants | 5 | 0

9. Secondary Outcome: Smoking Quit Attempts, as Measured by Number of Participant's Partners Who Reported One or Greater Quit Attempts
Time Frame: at the time of follow-up visit #2 (about 1 month post-intervention)
Population: For each arm, 12 partners reported current smoking at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 12 | 12
Participants | 2 | 1

10. Secondary Outcome: Smoking Quit Attempts, as Measured by Number of Other Household Members (Other Than the Participant or the Participant's Partner) Who Reported One or Greater Quit Attempts
Time Frame: at the time of follow-up visit #1 (about 2 weeks post-intervention)
Population: For the Motivational advice and free NRT arm, 7 household members (other than the participant or the participant's partner) reported current smoking at baseline. For the Motivational advice and free NRT arm, 6 household members (other than the participant or the participant's partner) reported current smoking at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

11. Secondary Outcome: Smoking Quit Attempts, as Measured by Number of Other Household Members (Other Than the Participant or the Participant's Partner) Who Reported One or Greater Quit Attempts
Time Frame: at the time of follow-up visit #2 (about 1 month post-intervention)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

12. Secondary Outcome: Home Smoking Ban Status, as Measured by Number of Participants Who Report a Home-smoking Ban.
Time Frame: From time of randomization to follow-up visit #2 (generally completed within 2-3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 16 | 16
Participants | 14 | 14

13. Secondary Outcome: Car Smoking Ban Status, as Measured by Number of Participants Who Report a Car-smoking Ban.
Time Frame: From time of randomization to follow-up visit #2 (generally completed within 2-3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
Number analyzed (Participants) | 16 | 16
Participants | 14 | 14

ADVERSE EVENTS:
Time Frame: 2-3 months
Arm/Group | Motivational Advice and Free NRT | Quitline Referral
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT04045964/Prot_SAP_000.pdf